CLINICAL TRIAL: NCT01056120
Title: Long Term Safety Profile of the PRO-Kinetic ENERGY Coronary Stent System in Daily Clinical Practice Multinational, Prospective, Non-randomized, Multi-centre, Non-interventional Trial
Brief Title: Long Term Safety Profile of the PRO-Kinetic ENERGY Coronary Stent System in Daily Clinical Practice
Acronym: ENERGY
Status: Completed | Type: Observational
Sponsor: Biotronik AG (Industry)
Responsible Party: Sponsor
Other Study IDs: C0903
Record Dates: First submitted 2010-01-25; First posted 2010-01-26 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2016-01

CONDITIONS: De Novo and Re-stenosed Coronary Artery Lesions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ENERGY-Population: Patient population in standard clinical care, according to the instructions for use and the inclusion / exclusion criteria. Registry patients should be enrolled consecutively to represent a typical set of patients at each site.
  The registry will collect clinical data from patients that have given their prior written consent. All data will be anonymized prior to data entry.
  Interventions: Device: Pro Kinetic Energy bare metal stent

INTERVENTIONS:
Device: Pro Kinetic Energy bare metal stent — PCI

SUMMARY:
To evaluate the clinical performance of the PRO-Kinetic ENERGY® coronary bare metal stent system in a patient population within that defined in the Instructions for Use.

ELIGIBILITY:
Inclusion Criteria:

* Patient signed informed consent for data release
* Patient eligible for percutaneous coronary intervention (PCI)
* De novo and re-stenosed coronary artery lesions
* Patient is geographically stable and willing to participate at all follow up assessments
* Patient is > 18 years of age

Exclusion Criteria:

* Patient receives more than one stent, which is not a PRO-Kinetic ENERGY stent within the same vessel
* Patient has a known allergy against aspirin, clopidogrel, ticlopidine, heparin or any other anticoagulation / antiplatelet therapy required for PCI
* Patient presents with ISR (in-stent restenosis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 1026 (Actual)
Dates: Start 2010-03; Primary Completion 2013-02 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
MACE (Cardiac death, clinically driven TLR, MI / AMI (STEMI / NSTEMI) | 6 months

SECONDARY OUTCOMES:
• MACE after 12 and 24 months • TVR after 6, 12 and 24 months • Stent Thrombosis at 6, 12 and 24 months acc. to the academic research consortium -ARC (13) | 6,12, 24 Months

CONTACTS AND LOCATIONS:
Overall Officials: Raimund Erbel, MD, Principal Investigator — Klinik für Kardiologie Westdeutsches Herzzentrum Essen, Universitätsklinikum Essen, Hufelandstrasse 55, D-45122 Essen, Germany
Locations (50):
- Austria (2):
  - Landeskrankenhaus Bruck an der Mur, Bruck an der Mur
  - Kardinal Schwarzenberg'sches Krankenhaus, Schwarzach Saint Veit
- Belgium (2):
  - Saint-Pierre University Hospital, Brussels
  - Cliniques Universitaires UCL de Mont-Godinne, Yvoir
- France (8):
  - Clinique Axium, Aix-en-Provence
  - Clinique Rhone Durance, Avignon
  - Clinique Convert, Bourg-en-Bresse
  - Centre Hospitalier de Chartres, Chartres
  - Clinique la Mutualiste, Grenoble
  - Clinique Générale de Marignane, Marignane
  - Centre Hospitalier de Pau, Pau
  - Clinique Saint Pierre, Perpignan
- Germany (17):
  - Westdeutsches Herzzentrum Essen, Essen, North Rhine-Westphalia
  - Herz- und Diabeteszentrum Nordrhein-Westfalen, Bad Oeynhausen
  - Charité-Universitätsm. Berlin Campus Charité-Mitte, Berlin
  - Vivantes Humboldt Klinikum, Berlin
  - Universitätsklinikum Bonn, Bonn
  - Klinikum Dortmund GmbH, Dortmund
  - Städ. Klinikum Dresden- Friedrichstadt, Dresden
  - Alfried Krupp Klinikum Essen, Essen
  - Vinzenz Krankenhaus, Essen
  - Asklepios Klinikum St. Georg, Hamburg
  - St. Marien Hospital, Lünen
  - Niels-Stensen-Kliniken Marienhospital Osnabrück, Osnabrück
  - Universitätsklinikum Regensburg, Regensburg
  - Diakonissen-Stiftungs-Krankenhaus Speyer, Speyer
  - Elbe Klinikum Stade GmbH, Stade
  - SRH Zentralklinikum Suhl, Suhl
  - Marien-Hospital Witten GmbH, Witten
- Craigavon Cardiac Centre, Craigavon, Ireland
- Israel (5):
  - Assaf Harofeh Medical Center, Beer Yakov
  - Carmel Medical Center, Haifa
  - Rambam Medical Center, Haifa
  - Kaplan Medical Center, Rehovot
  - Ziv Medical Center, Safed
- Latvia (2):
  - Pauls Stradins Clinical University Hospital, Riga
  - Riga East Clinical University Hospital, Riga
- Netherlands (3):
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - VU Medisch Centrum, Amsterdam
  - Academisch Ziekenhuis Maastricht, Maastricht
- Spain (7):
  - Hospital Torrecardenas, Almería
  - Hospital Clinic I Provinvial de Barcelona, Barcelona
  - Hospital de la Santa Creu i San Pau, Barcelona
  - Hospital San Pedro de Alcantara, Cáceres
  - Hospital de Puerta de Hierro, Madrid
  - Hospital Mexoeiro, Vigo
  - Hospital Galdakao, Vizcaya
- Switzerland (3):
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Clinique Cecil, Lausanne
  - University Hospital Zürich, Zurich

REFERENCES:
- [Derived] Scheinert D, Schulte KL, Zeller T, Lammer J, Tepe G. Paclitaxel-releasing balloon in femoropopliteal lesions using a BTHC excipient: twelve-month results from the BIOLUX P-I randomized trial. J Endovasc Ther. 2015 Feb;22(1):14-21. doi: 10.1177/1526602814564383. PMID 25775674
- [Derived] Erbel R, Eggebrecht H, Roguin A, Schroeder E, Philipp S, Heitzer T, Schwacke H, Ayzenberg O, Serra A, Delarche N, Luchner A, Slagboom T; ENERGY Investigators. Prospective, multi-center evaluation of a silicon carbide coated cobalt chromium bare metal stent for percutaneous coronary interventions: two-year results of the ENERGY Registry. Cardiovasc Revasc Med. 2014 Nov-Dec;15(8):381-7. doi: 10.1016/j.carrev.2014.10.002. Epub 2014 Oct 15. PMID 25456414